CLINICAL TRIAL: NCT02219308
Title: Pain Control for Intrauterine Device Placement: A Randomized Controlled Trial of Paracervical Block
Brief Title: Pain Control for Intrauterine Device Placement Using Paracervical Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Women's Reproductive Health Research (K12) Scholar, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141025
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pain Due to Intrauterine Contraceptive Device
Keywords: Contraception; Pain; Intrauterine Device; Paracervical Block
MeSH Terms: conditions — Pain | interventions — Anesthesia, Obstetrical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracervical Block (PCB) (Experimental): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, where tenaculum will be placed.
  Subject then receives paracervical block of 18 mL 1% buffered Lidocaine. Provider then places IUD.
  Interventions: Procedure: Paracervical Block (PCB)
- No Paracervical Block (Sham PCB) (Sham Comparator): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, where tenaculum will be placed.
  Subject then receives Sham paracervical block with capped needle. Provider then places IUD.
  Interventions: Procedure: No Paracervical Block (Sham PCB)

INTERVENTIONS:
Procedure: Paracervical Block (PCB) — Drug: 1% Lidocaine Hydrochloride
  Injection of 2 mL 1% buffered lidocaine solution at anterior lip of cervix and 18 mL 1% buffered lidocaine solution evenly distributed between 4 o'clock and 8 o'clock positions of cervix with standard 22 gauge spinal needle.
  IUD placement then proceeds
  Arms: Paracervical Block (PCB)
Procedure: No Paracervical Block (Sham PCB) — Drug: 1% Lidocaine Hydrochloride
  Injection of 2 mL 1% buffered lidocaine solution at anterior lip of cervix with standard 22 gauge spinal needle. Capped spinal needle is then held against the cervix at 4 o'clock and 8 o'clock positions of cervix, lightly so as not to cause blanching, indentation, or pain.
  IUD placement then proceeds
  Arms: No Paracervical Block (Sham PCB)

SUMMARY:
Intrauterine device (IUD) placement can be painful for patients during and after the procedure. Fear of pain from IUD insertion can be a barrier to obtaining this highly effective long acting reversible contraception. Currently there are no proven effective methods for reduction of pain during and after placement of modern IUDs. Paracervical block pain may decrease this placement pain.

DETAILED DESCRIPTION:
Modern IUDs are highly effective long acting reversible forms of contraception. The Mirena IUD is 99.8% effective and the Paragard copper IUD is 99.2% effective in preventing pregnancy. Fear of IUD placement can be a barrier to obtaining this highly effective form of birth control. The current standard of care for pain management during and after IUD placement is no medication, as randomized control trials published to date have limited data regarding use of medications to decrease pain. There has been one trial to suggest that the use of naproxen with 1% lidocaine paracervical block (PCB) compared to PCB alone may decrease pain after IUD placement in primarily nulliparous patients. However, this study was with the much wider and no longer available Dalkon Shield IUD. In addition, this study did not show any significant decrease in pain scores during IUD placement. Studies to evaluate effectiveness of ibuprofen and misoprostol have shown no significant decrease in pain scores during and after IUD insertion, although the majority of participants in these studies were multiparous. There is some suggestion that 2% lidocaine gel one minute prior to IUD insertion may have some decrease in pain, although this study was poorly designed.

Although there is no standard of care in regards to pain medication administration prior to IUD placement, providers often suggest paracervical prior IUD insertion among nulliparous women. Therefore the primary aim of this study is to determine whether a paracervical block (PCB) decreases pain associated with intrauterine device (IUD) placement compared to no paracervical block. We hypothesize that administration of a PCB of 20 mL 1% buffered lidocaine prior to IUD placement will decrease pain scores by at least 20mm on a visual analog scale at various time points during IUD placement when compared to no paracervical block.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* English or Spanish speaking
* Present for intrauterine device placement for contraception or menorrhagia (in the case of Mirena IUD insertion).

Exclusion Criteria:

* Pregnancy
* Any diagnosed chronic pain issues (i.e. fibromyalgia, endometriosis, dysmenorrhea, irritable bowel syndrome, interstitial cystitis)
* If the patient has taken any pain medications within 6 hours of enrollment, including aspirin or other NSAIDs
* Misoprostol administration within 24 hours of enrollment
* History of prior IUD insertion
* Known contraindications to IUD

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD MPH, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - UCSD, San Diego, California
  - Planned Parenthood Mission Bay Parker Center, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RH, Bartz D, Grimes DA, Hubacher D, O'Brien P. Interventions for pain with intrauterine device insertion. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007373. doi: 10.1002/14651858.CD007373.pub2. PMID 19588429
- [Background] Cetin A, Cetin M. Effect of deep injections of local anesthetics and basal dilatation of cervix in management of pain during legal abortions. A randomized, controlled study. Contraception. 1997 Aug;56(2):85-7. doi: 10.1016/s0010-7824(97)00096-6. PMID 9315416
- [Background] Edelman AB, Schaefer E, Olson A, Van Houten L, Bednarek P, Leclair C, Jensen JT. Effects of prophylactic misoprostol administration prior to intrauterine device insertion in nulliparous women. Contraception. 2011 Sep;84(3):234-9. doi: 10.1016/j.contraception.2011.01.016. Epub 2011 Mar 3. PMID 21843686
- [Background] Hubacher D, Reyes V, Lillo S, Zepeda A, Chen PL, Croxatto H. Pain from copper intrauterine device insertion: randomized trial of prophylactic ibuprofen. Am J Obstet Gynecol. 2006 Nov;195(5):1272-7. doi: 10.1016/j.ajog.2006.08.022. PMID 17074548
- [Background] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115
- [Background] Massey SE, Varady JC, Henzl MR. Pain relief with naproxen following insertion of an intrauterine device. J Reprod Med. 1974 Dec;13(6):226-31. No abstract available. PMID 4612152
- [Background] Mosher WD, Jones J. Use of contraception in the United States: 1982-2008. Vital Health Stat 23. 2010 Aug;(29):1-44. PMID 20939159
- [Background] O'Connell K, Jones HE, Simon M, Saporta V, Paul M, Lichtenberg ES; National Abortion Federation Members. First-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2009 May;79(5):385-92. doi: 10.1016/j.contraception.2008.11.005. Epub 2008 Dec 11. PMID 19341852
- [Background] Phair N, Jensen JT, Nichols MD. Paracervical block and elective abortion: the effect on pain of waiting between injection and procedure. Am J Obstet Gynecol. 2002 Jun;186(6):1304-7. doi: 10.1067/mob.2002.123734. PMID 12066113
- [Background] Rabin JM, Spitzer M, Dwyer AT, Kaiser IH. Topical anesthesia for gynecologic procedures. Obstet Gynecol. 1989 Jun;73(6):1040-4. doi: 10.1097/00006250-198906000-00027. PMID 2657523
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman A. Pain control in first trimester surgical abortion. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD006712. doi: 10.1002/14651858.CD006712.pub2. PMID 19370649
- [Background] Roche NE, Li D, James D, Fechner A, Tilak V. The effect of perioperative ketorolac on pain control in pregnancy termination. Contraception. 2012 Mar;85(3):299-303. doi: 10.1016/j.contraception.2011.10.001. Epub 2011 Nov 30. PMID 22133656
- [Background] Wiebe ER, Rawling M. Pain control in abortion. Int J Gynaecol Obstet. 1995 Jul;50(1):41-6. doi: 10.1016/0020-7292(95)02416-a. PMID 7556858
- [Background] Wiebe ER. Comparison of the efficacy of different local anesthetics and techniques of local anesthesia in therapeutic abortions. Am J Obstet Gynecol. 1992 Jul;167(1):131-4. doi: 10.1016/s0002-9378(11)91645-7. PMID 1442914
- [Background] Zieman, Mimi et al. A Pocket Guide to Managing Contraception. The Bridging Gap Foundation. © 2010
- [Background] Zullo F, Pellicano M, Stigliano CM, Di Carlo C, Fabrizio A, Nappi C. Topical anesthesia for office hysteroscopy. A prospective, randomized study comparing two modalities. J Reprod Med. 1999 Oct;44(10):865-9. PMID 10554747
- [Derived] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion: Nulliparous women, 18-45, requesting IUD, seen in our clinic from October 2014 through October 2017 Exclusion: pregnancy, diagnosed chronic pain issues, use of pain medication within 6 hours, misoprostol administration within 24 hours, history of prior IUD placement, known contraindications to IUD placement.
Groups:
- No Paracervical Block (Sham PCB): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, then receives Sham paracervical block with capped needle.
- Paracervical Block (PCB): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, then receives paracervical block of 18 mL 1% buffered Lidocaine.
Period: Overall Study
Arm/Group | No Paracervical Block (Sham PCB) | Paracervical Block (PCB)
Started | 32 | 35
Completed | 31 | 33
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- No Paracervical Block (Sham PCB): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, where tenaculum will be placed.
  Subject then receives Sham paracervical block with capped needle. Provider then places IUD.
  No Paracervical Block (Sham PCB): Drug: 1% Lidocaine Hydrochloride
  Injection of 2 mL 1% buffered lidocaine solution at anterior lip of cervix with standard 22 gauge spinal needle. Capped spinal needle is then held against the cervix at 4 o'clock and 8 o'clock positions of cervix, lightly so as not to cause blanching, indentation, or pain.
  IUD placement then proceeds
- Paracervical Block (PCB): Subject receives 2 mL 1% buffered Lidocaine anesthetic at anterior lip of cervix, where tenaculum will be placed.
  Subject then receives paracervical block of 18 mL 1% buffered Lidocaine. Provider then places IUD.
  Paracervical Block (PCB): Drug: 1% Lidocaine Hydrochloride
  Injection of 2 mL 1% buffered lidocaine solution at anterior lip of cervix and 18 mL 1% buffered lidocaine solution evenly distributed between 4 o'clock and 8 o'clock positions of cervix with standard 22 gauge spinal needle.
  IUD placement then proceeds
- Total: Total of all reporting groups
Arm/Group | No Paracervical Block (Sham PCB) | Paracervical Block (PCB) | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (3.4) | 26.1 (3.9) | 25.45 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 21 | 41
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Pain With Intrauterine Device (IUD) Placement
Description: Distance (mm) from the left of the 100-mm visual analog scale (reflecting magnitude of pain) recorded at time of IUD Placement. Scale range is from 0mm (no pain) to 100mm (worst pain possible). A lower score (less pain) is considered a better outcome.
Time Frame: Moment of IUD insertion
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | No Paracervical Block (Sham PCB) | Paracervical Block (PCB)
Number analyzed (Participants) | 31 | 33
mm | 54 [33 to 75] | 33 [10 to 56]

2. Secondary Outcome: Median Pain Scores for All Time Points
Description: Distance (mm) from the left of the 100-mm visual analog scale of pain at various time points. Scale range is 0mm (no pain) to 100mm (worst pain possible). Lower scores are considered better outcomes.
Time Frame: Anticipation of procedure through 5 minutes after IUD placement
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | No Paracervical Block (Sham PCB) | Paracervical Block (PCB)
Number analyzed (Participants) | 31 | 33
mm
  Anticipated Pain | 51 [30 to 70] | 58 [48 to 68]
  Baseline Pain | 0 [0 to 2] | 0 [0 to 2]
  Speculum Insertion | 6 [2 to 20] | 10 [4 to 14]
  Capped Needle or PCB | 8 [2 to 20] | 30 [17 to 47]
  Tenaculum placement | 10 [4 to 19] | 15 [6 to 24]
  Uterine Sounding | 47 [24 to 65] | 30 [8 to 43]
  IUD placement | 54 [33 to 75] | 33 [10 to 56]
  5 mins after IUD placement | 27 [15 to 50] | 12 [6 to 27]
  Overall pain | 51 [21 to 65] | 30 [16 to 48]

ADVERSE EVENTS:
Time Frame: IUD insertion procedure: from anticipation of procedure through 5 minutes after IUD placement. Total time approximately 20 minutes.
Arm/Group | No Paracervical Block (Sham PCB) | Paracervical Block (PCB)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02219308/Prot_SAP_000.pdf